CLINICAL TRIAL: NCT00421473
Title: Drug Interactions Between ATOvaquone Used in MAlaria Prophylaxis and Antiretroviral Agents in HIV-1 Infected Patients (ATOMA)
Brief Title: Drug Interaction Study Between Atovaquone and Antiretroviral Agents in HIV-1 Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UMCN-AKF 06.02
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; Malaria
Keywords: HIV; Malaria prophylaxis; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Malaria | interventions — atovaquone, proguanil drug combination

INTERVENTIONS:
Drug: Atovaquone / Proguanil

SUMMARY:
Malarone® (atovaquone/proguanil) is frequently used in malaria prophylaxis. Unfortunately, there are indications that certain anti-HIV agents may decrease atovaquone plasma levels by induction of atovaquone metabolism.

For travelling HIV patients, the clinical consequences of these possible drug drug interactions are serious, since a diminished exposure to the anti-malarial drug will result in suboptimal prophylaxis of malaria and potential development of drug resistant strains of Plasmodium falciparum.

The purpose of this study is to find out if HIV patients using HAART regimes with either lopinavir/ritonavir, atazanavir/ritonavir or efavirenz have lower atovaquone plasma levels than healthy volunteers after a single dose of atovaquone/proguanil.

ELIGIBILITY:
Inclusion Criteria:

For healthy volunteers

* 18 - 65 years
* smoking habits < 10 cigarettes, 2 cigars or 2 pipes
* BMI between 18 and 30 kg/m2
* able and willing to sign informed consent form
* subject is in a good age-appropriate health condition
* subject has a normal blood pressure and pulse rate

For HIV patients

* HIV-infected as documented by positive HIV antibody test and confirmed by Western Blot.
* CD4+ > 200 * 10E6 per Liter.
* 18 - 65 years
* BMI between 18 and 30 kg/m2
* able and willing to sign informed consent form
* use of lopinavir/ritonavir, atazanavir/ritonavir or efavirenz for at least 1 month in a dose of 400/100mg bid, 300/100 mg QD, or 600 mg QD respectively

Exclusion Criteria healthy volunteers:

* History of sensitivity/idiosyncrasy to atovaquone/proguanil or chemically related compounds or excipients.
* Positive HIV test.
* Positive HbsAg test (hepatitis B) or positive hepatitis C test.
* Therapy with any drug (for two weeks preceding dosing), except for paracetamol.
* Creatinine clearance < 60 mL/min (calculated from serum creatinine)
* Current diarrhoea.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose.
* Donation of blood within 60 days prior to the first dose.
* Pregnant female (as confirmed by an HCG test performed less than 3 weeks before the first dose) or breast-feeding female.
* Abnormal serum transaminases, determined as levels being > 3 times up-per limit of normal
* Febrile illness within 3 days before the first dose

Exclusion criteria HIV patients:

* History of sensitivity/idiosyncrasy to atovaquone/proguanil or chemically related compounds or excipients.
* Suspicion of non-adherence to the HIV medication.
* Current diarrhoea.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* Inability to understand the nature and extent of the trial and the procedures required.
* Pregnant female (as confirmed by an HCG test performed less than 3 weeks before the first dose) or breast-feeding female.
* Abnormal serum transaminases determined as levels being > 3 times upper limit of normal
* Creatinine clearance < 60 mL/min (calculated from serum creatinine).
* Any change in antiretroviral medication within 1 month immediately pre- ceding the dose of atovaquone/proguanil.
* Concomitant use of medications that interfere with atovaquone or proguanil pharmacokinetics: anti-coagulants, aurothioglucose, chloroquine, cimetidine, fluoxetine, fluvoxamine, metoclopramide, omeprazole, magnesiumtrisilicate, rifabutin, rifampin, tetracycline, typhoid vaccine, topiramate.
* Use of a HAART regime containing both lopinavir/ritonavir and another protease inhibitor or a NNRTI.
* Use of a HAART regime containing both atazanavir/ritonavir and another protease inhibitor or a NNRTI.
* Use of a HAART regime containing both efavirenz and one or more protease inhibitors or nevirapine.
* Active hepatobiliary or hepatic disease
* Alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic blood samples will be taken just before dosing Malarone, and 12 samples in the time between 0,5 hour and 168 hours after dosing.

SECONDARY OUTCOMES:
Blood will be taken for genotyping of CYP2C19 at study day 1.
HIV-1 RNA and CD4 determination will be done (HIV patients only) at inclusion screening

CONTACTS AND LOCATIONS:
Overall Officials: D.M. Burger, Dr., Principal Investigator — Radboud University Medical Centre Nijmegen
Locations (5):
- Netherlands (5):
  - Alysis Zorggroep loc. Rijnstate, Arnhem, Gelderland
  - Radboud University Medical Centre Nijmegen, Nijmegen, Gelderland
  - Elisabeth hospital, Tilburg, North Brabant
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland

REFERENCES:
- [Result] van Luin M, Van der Ende ME, Richter C, Visser M, Faraj D, Van der Ven A, Gelinck L, Kroon F, Wit FW, Van Schaik RH, Kuks PF, Burger DM. Lower atovaquone/proguanil concentrations in patients taking efavirenz, lopinavir/ritonavir or atazanavir/ritonavir. AIDS. 2010 May 15;24(8):1223-6. doi: 10.1097/QAD.0b013e3283389129. PMID 20299957